CLINICAL TRIAL: NCT00473616
Title: A Phase I Open-label, Multi-center, Dose-escalation and Safety Expansion Study to Assess Safety, Tolerability, and Pharmacokinectics of AZD7762 Administered as a Single Intravenous Agent and in Combination With Weekly Standard Dose of Irinotecan in Patients With Advanced Solid Malignancies.
Brief Title: Phase I Single Ascending Dose/Multiple Ascending Dose in Patients Treated With AZD7762 and Irinotecan
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination of the study was made after a full review of program data and assessment of the current risk-benefit profile.
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1040C00004
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Advanced Solid Tumors; Cancer; Advanced Solid Malignancies
Keywords: Phase I; solid tumors; solid malignancies; cancer Eligibility
MeSH Terms: conditions — Neoplasms | interventions — 3-(carbamoylamino)-5-(3-fluorophenyl)-N-(3-piperidyl)thiophene-2-carboxamide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD7762 monotherapy followed by AZD7762 + irinotecan
  Interventions: Drug: AZD7762; Drug: Irinotecan

INTERVENTIONS:
Drug: AZD7762 — intravenous infusion
Drug: Irinotecan — intravenous injection
  Other Names: Campto®; Camptosar®; irinotecan hydrochloride

SUMMARY:
This is an open-label, multi-center, dose-escalation and safety expansion, Phase I study to evaluate the safety, tolerability, and pharmacokinectics and to investigate biomarker changes of AZD7762 administered as a single intravenous unit and in combination with irinotecan. The study is sponsored by AstraZeneca.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors for which standard treatment doesn't exist or is no longer effective.
* Must be suitable for treatment with irinotecan
* Relatively good overall health other than your cancer

Exclusion Criteria:

* Poor bone marrow function (not producing enough blood cells)
* Serious heart conditions
* Poor liver or kidney function
* Any prior anthracycline treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the safety and tolerability of AZD7762 alone and in combination with Irinotecan | assessed after each course of treatment

SECONDARY OUTCOMES:
To determine the single-dose (after the first single-agent dose) and combination-dose (afer the 2nd combination dose) pharmacokinetics (PK) of AZD7762. | assessed after each course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — AstraZeneca
Locations (3):
- United States (3):
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research site, Nashville, Tennessee